CLINICAL TRIAL: NCT05967065
Title: Diagnostic Precision Study on Vibration Induced Nystagmus Test for SCDS by Ortofone
Brief Title: Diagnostic Precision Study on Vibration Induced Nystagmus Test for SCDS by Ortofone B250 Skull Vibration Protocol
Acronym: VIN by B250
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical issues in testing procedure
Sponsor: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Luca Verrecchia, Principal investigator, Region Stockholm
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RegionStockholm
Record Dates: First submitted 2023-06-01; First posted 2023-08-01 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Superior Canal Dehiscence Syndrome; Vestibular Disorder
MeSH Terms: conditions — Semicircular Canal Dehiscence; Vestibular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular disorders (Other): Patients uppfilling vestibular disorders diagnostic criterias
  Interventions: Diagnostic Test: vibration induced nystagmus test
- healthy control subjects (Other): Patients without past or ongoing vestibular or balance disorders
  Interventions: Diagnostic Test: vibration induced nystagmus test

INTERVENTIONS:
Diagnostic Test: vibration induced nystagmus test — Vibration induced nystagmus test by bone transducer B250.

SUMMARY:
to study the videonystagmography response to a bone conducted vibration on the mastoid by B250 bone transducer in patients affected by vestibular loss, Menieres disease and Superior Semicircular Canal Dehiscence Syndrome vs healthy control subjects

ELIGIBILITY:
Inclusion Criteria:

Patients affected by certain vestibular disorders.

Exclusion Criteria:

Patients with vertigo and dizziness without certain diagnosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
measure of eye movements | through study completion, an average of 18 months
  angular velocity of eye movements during skull vibration.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Hearing and Balance Unit, Stockholm, Sweden